CLINICAL TRIAL: NCT00156858
Title: Busulfan and Fludarabine as Conditioning for Allogeneic Stem Cell
Brief Title: Busulfan and Fludarabine as Conditioning for Allogeneic Stem Cell Transplantation: a Pharmacokinetic Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10156; 717905172
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-09

CONDITIONS: Hematologic Malignancy
Keywords: pharmacokinetics; transplantation; busulfan
MeSH Terms: conditions — Hematologic Neoplasms

INTERVENTIONS:
Drug: intravenous busulfan

SUMMARY:
A study of pharmacokinetics of daily intravenous busulfan

DETAILED DESCRIPTION:
A study of pharmacokinetics of daily intravenous busulfan

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing transplantation

Exclusion Criteria:

-

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1998-01; Study Completion 2010-12

PRIMARY OUTCOMES:
pharmacokinetic data

CONTACTS AND LOCATIONS:
Overall Officials: James Russell, FRCp, Principal Investigator — Alberta Cancerboard
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada